CLINICAL TRIAL: NCT00611013
Title: Magnetic Resonance Imaging and Spectroscopy at High Field
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Min-Ying (Lydia) Su, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UCI-HS-2002-2611
Record Dates: First submitted 2008-01-12; First posted 2008-02-08 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Development of multi-purpose novel imaging protocols
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Some participants may receive MRI contrast agent, 0.1 mmol/kg

SUMMARY:
Evaluating novel MR imaging techniques on volunteers.

DETAILED DESCRIPTION:
The aim of this study is twofold. The first aim is to evaluate new MRI techniques developed by the investigators of this protocol on human volunteers. The second aim is to assist other investigators who need to use MR images obtained on this device for their own research. MR images and/or spectroscopy data will be acquired from the participants in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal volunteers for imaging protocol optimization.

Exclusion Criteria:

* Patients with implanted surgical clips (hemostatic clips) or other ferromagnetic material,
* Patients engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or who may have imbedded metal fragments from military activities,
* Patients with permanent (tattoo) eye-liner or with facial make-up (severe eye irritation has been reported),
* Patients with compromised thermoregulatory systems (e.g. certain cancer patients),
* Patients with metallic implants, because they may cause artifacts in diagnostic images due to magnetic field distortion,
* Patients with implanted prosthetic heart valves,
* Patients with pacemakers, neuro-stimulation devices,
* Pregnant patients (the safety of magnetic resonance examination has not been completely established for embryos and fetuses),
* Subjects who have received orthodontic work involving ferromagnetic materials,
* Subjects who have claustrophobia, and
* The patients unwilling to participate in the study or fail to sign the consent form.
* Subjects who are pregnant or breast-feeding will be excluded from the contrast enhanced MRI studies.
* Subjects who had allergic response to contrast agents previously will be excluded from contrast enhanced MRI studies.
* Subjects with known history of asthma, allergic conditions, severe renal insufficiency, sickle cell anemia, chronic hemolytic anemia, gastrointestinal disorders will also be excluded from contrast enhanced MRI studies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-06; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
General purpose novel magnetic resonance imaging contrasts, developments for improved magnetic resonance image quality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lutfi T Muftuler, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- Center for Functional Onco-Imaging, University of California, Irvine, California, United States